CLINICAL TRIAL: NCT06448351
Title: Manipulating E-Cigarette Nicotine to Promote Public Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Theodore Wagener, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: OSU-23143; NCI-2023-05712 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-05-22; First posted 2024-06-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Specimen Handling; Carbon Monoxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Personnel performing the assays will be blinded to the status of the sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (28):
- Phase 1, Arm 1 (High, Nic, S) (Experimental): Participants are randomized to vape one out of the eight study e-liquids in a 10-puff vaping session over 5 minutes using the e-cig study device and then in an ad libitum puffing session over 60 minutes. The 8 e-liquids vary in nicotine concentration (low [20 mg/g] or high [50 mg/g]), form (Nic or NicH+), and isomer (S-nicotine or R/S nicotine).
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 1, Arm 2 (High, Nic, R/S) (Experimental): Participants are randomized to vape one out of the eight study e-liquids in a 10-puff vaping session over 5 minutes using the e-cig study device and then in an ad libitum puffing session over 60 minutes. The 8 e-liquids vary in nicotine concentration (low [20 mg/g] or high [50 mg/g]), form (Nic or NicH+), and isomer (S-nicotine or R/S nicotine).
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 1, Arm 3 (Low, Nic, S) (Experimental): Participants are randomized to vape one out of the eight study e-liquids in a 10-puff vaping session over 5 minutes using the e-cig study device and then in an ad libitum puffing session over 60 minutes. The 8 e-liquids vary in nicotine concentration (low [20 mg/g] or high [50 mg/g]), form (Nic or NicH+), and isomer (S-nicotine or R/S nicotine).
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 1, Arm 4 (Low, Nic, R/S) (Experimental): Participants are randomized to vape one out of the eight study e-liquids in a 10-puff vaping session over 5 minutes using the e-cig study device and then in an ad libitum puffing session over 60 minutes. The 8 e-liquids vary in nicotine concentration (low [20 mg/g] or high [50 mg/g]), form (Nic or NicH+), and isomer (S-nicotine or R/S nicotine).
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 1, Arm 5 (High, NicH+, S) (Experimental): Participants are randomized to vape one out of the eight study e-liquids in a 10-puff vaping session over 5 minutes using the e-cig study device and then in an ad libitum puffing session over 60 minutes. The 8 e-liquids vary in nicotine concentration (low [20 mg/g] or high [50 mg/g]), form (Nic or NicH+), and isomer (S-nicotine or R/S nicotine).
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 1, Arm 6 (High, NicH+, R/S) (Experimental): Participants are randomized to vape one out of the eight study e-liquids in a 10-puff vaping session over 5 minutes using the e-cig study device and then in an ad libitum puffing session over 60 minutes. The 8 e-liquids vary in nicotine concentration (low [20 mg/g] or high [50 mg/g]), form (Nic or NicH+), and isomer (S-nicotine or R/S nicotine).
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 1, Arm 7 (Low, NicH+, S) (Experimental): Participants are randomized to vape one out of the eight study e-liquids in a 10-puff vaping session over 5 minutes using the e-cig study device and then in an ad libitum puffing session over 60 minutes. The 8 e-liquids vary in nicotine concentration (low [20 mg/g] or high [50 mg/g]), form (Nic or NicH+), and isomer (S-nicotine or R/S nicotine).
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 1, Arm 8 (Low, NicH+, R/S) (Experimental): Participants are randomized to vape one out of the eight study e-liquids in a 10-puff vaping session over 5 minutes using the e-cig study device and then in an ad libitum puffing session over 60 minutes. The 8 e-liquids vary in nicotine concentration (low [20 mg/g] or high [50 mg/g]), form (Nic or NicH+), and isomer (S-nicotine or R/S nicotine).
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 1 (High, 5%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 2 (High, 5%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 3 (Low, 5%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 4 (Low, 5%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 5 (High, 25%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 6 (High, 25%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 7 (Low, 25%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 8 (Low, 25%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 9 (High, 45%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 10 (High, 45%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 11 (Low, 45%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 12 (Low, 45%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 13 (High , 65%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 14 (High , 65%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 15 (Low, 65%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 16 (Low, 65%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 17 (High, 85%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 18 (High, 85%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 19 (Low, 85%, S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration
- Phase 2, Arm 20 (Low, 85%, R/S) (Experimental): Participants vape 20 different study e-liquids varying in concentration (low [20 mg/g] or high [50 mg/g]), freebase nicotine percentage (5%, 25%, 45%, 65%, or 85%), and isomer (S-nicotine or R/S nicotine) using the e-cig study device during two visits.
  Interventions: Procedure: Biospecimen Collection; Procedure: Carbon Monoxide Measurement; Other: Vaping session; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Carbon Monoxide Measurement — Undergo CO test
  Other Names: Carbon Monoxide; CMONOX
Other: Vaping session — Sample study e-liquids in vaping sessions at research lab with e-cig study device
  Other Names: Vaping e-liquid
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial explores the manipulation of e-cigarette (EC) nicotine to promote public health. Researchers are trying to understand and gather information about how the strength, form, and structure of nicotine in products play a significant role in their potential for addiction and how they might affect health risks. The information gained from this study may allow researchers to understand how these aspects of nicotine influence the potential for addiction, how people puff on ECs, how the body processes nicotine, and any potential harmful effects it might have on health. Exploring these specific characteristics of nicotine may also determine if an EC product standard could help identify optimal nicotine levels for users.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the pharmacological, metabolic, and behavioral impact of nicotine dimensions. (Study 1) II. Assess the toxicity resulting from different nicotine dimension combinations. (Study 1) III. Across ecologically valid nicotine concentrations and isomer ratios, determine free-base (FB) nicotine fractions with minimal appeal to young adult EC users but sufficient appeal to smokers. (Study 2)

OUTLINE:

Phase 1 (STUDY 1): Participants are randomized to the order of 8 e-liquid combinations varying in nicotine concentration, form, and isomer.

Participants participate in a 10-puff vaping session over 5 minutes with a study e-liquid using the study EC device followed by a 60 minute washout period and then an ad libitum puffing session over 60 minutes at each lab visit. Patients are also given a new pre-filled study device corresponding to the study e-liquid they will use for the subsequent visit to practice at home. Puffing sessions continue with a new study e-liquid at each of the 8 lab visits lasting up to 4 hours each. Participants also undergo carbon monoxide (CO) testing and blood and urine sample collection on study.

Phase 2 (STUDY 2): Participants are randomized to the order of 20 e-liquid combinations varying in concentration, FB fractions, and isomer.

Participants will take part in a 2-puff vaping session with each of the 20 study e-liquids using the study EC device with a 20-minute washout period between each vaping session. Vaping sessions are grouped into two visits, each lasting up to 5 hours and consisting of 10 e-liquids. Participants also undergo CO testing and blood and urine sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* Current exclusive young adult EC user for at least the past 3 months (confirmed by cotinine testing strip) between 21-24 years old with no/minimal history of smoking cigarettes (≤ 10 cigarettes in entire life)
* Current older adult smoker (daily use, ≥ 100 cigarettes in entire life) aged 25-65 with interest in trying an EC
* Willing to abstain from all nicotine, tobacco products, and marijuana for at least 12 hours before study visits
* Read and speak English

Exclusion Criteria:

* Currently attempting to quit nicotine or tobacco products
* Currently pregnant (will be verified with urine pregnancy test), planning to become pregnant, or breastfeeding
* If age 21-24 years old AND use of any tobacco products other than ECs (use of >10 cigarettes in entire life; use of >10 traditional cigars, cigarillos, or filtered cigars in entire life; use of smokeless tobacco products >10 times in entire life; or hookah in the last 30 days).
* Self-reported diagnosis of lung disease including asthma, cystic fibrosis, or chronic obstructive pulmonary disease
* New or unstable cardiovascular disease diagnosed within the past 3 months
* Use of medications that are inducers of CYP2A6 enzyme such as rifampicin, dexamethasone, phenobarbital, and other anti-convulsion drugs

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Nicotine pharmacokinetics: Maximum nicotine blood level (Cmax) (Study 1) | Immediately before puffing (-5 minutes), and at 5, 15, 60, and 120 minutes after the start of the puffing session
  Blood nicotine samples will be assayed using liquid chromatography tandem mass spectrometry (LC-MS/MS) with deuterated internal standards.
Nicotine pharmacokinetics: Time to maximum blood level (Tmax) (Study 1) | Immediately before puffing (-5 minutes), and at 5, 15, 60, and 120 minutes after the start of the puffing session
  Blood nicotine samples will be assayed using LC-MS/MS with deuterated internal standards.
Nicotine pharmacokinetics: Area under the curve (AUC) (Study 1) | Immediately before puffing (-5 minutes), and at 5, 15, 60, and 120 minutes after the start of the puffing session
  Blood nicotine samples will be assayed using LC-MS/MS with deuterated internal standards.
Nicotine metabolism (Study 1) | At 60 minutes after the start of each puffing session
  The rate of nicotine metabolism will be assessed using the standard method of nicotine metabolite ration (NMR) = hydroxycotinine/cotinine, modified to reflect stereoselective metabolism. Plasma concentration of cotinine, and hydroxycotinine will be measured by chiral LC-MS/MS based on previous methods and quantified using the ratio of metabolites to internal standards.
Reactive oxygen species (ROS) (Study 1) | Up to 2 years
  The recorded puffing topographies will be sent to the analytical lab for "puff playback" generation of EC aerosols and quantification of ROS. We will use an acellular ROS assay previously developed by our team as a generic toxicity assessment method.
Nicotine toxicity measures (Study 1) | Up to 2 years
  Will be assessed by carbonyl yields reported as ug/session or ug/puff or normalized per nicotine yield for a head-to-head comparison between different nicotine conditions.
In vitro nicotine toxicity measures: Cell cycle and proliferation (Study 1) | Up to 2 years
  Will be assessed by cell cycle and proliferationg.
In vitro nicotine toxicity measures: Cytotoxicity (Study 1) | Up to 2 years
  Will be assessed by cytotoxicity, senescence.
In vitro nicotine toxicity measures: Senescence (Study 1) | Up to 2 years
  Will be assessed by senescence.
In vitro nicotine toxicity measures: RNA sequencing (Study 1) | Up to 2 years
  Will be assessed by RNA sequencing.
Nicotine yield (Study 1) | Up to 2 years
  Using a dilute-and-shoot method developed by our team, nicotine yield in EC aerosol will be quantified using the "playback" technique (i.e., use topography collected from participants to machine-generate EC aerosols) and GC-MS method, developed by our group to minimize the PG/VG interference not addressed by other methods.
Modified Cigarette Evaluation Questionnaire (mCEQ)(Study 1) | Study visits 2 through 9
  The modified Cigarette Evaluation Questionnaire (mCEQ) will assess subjective responses. The 11-item mCEQ includes five subscales: Smoking Satisfaction, Psychological Reward, Aversion, Enjoyment of Respiratory Tract Sensations, and Craving Reduction, with items rated from 1 (not at all) to 7 (extremely likely). Items are averaged to create each of the subscales also ranging from 1 to 7 with higher values indicating greater levels of smoking satisfaction, psychological reward, aversion, enjoyment of respiratory tract sensations, and craving reduction.
Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form (QSU) | Study visits 2 through 9
  Smoking and vaping urges/craving will be measured using the Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form with a modified version (replacing the word "cigarette" with "e-cigarette") for EC users. This is a 10-item measure where participants rate smoking/vaping-related items on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Similar to previous studies, we will collapse the items into two previously identified factors (Factor 1: strong desire and intention to smoke/vape; Factor 2: anticipation of relief from withdrawal symptoms). Scores are calculated by summing the items and range from 5 to 35 for each of the factors with higher scores indicating greater craving to smoke/vape.
Drug Effects/Liking Questionnaire (DEQ)(Study 1) | Study visits 2 through 9
  Assess the desire and liking of products, positive and negative effects (i.e., side effects), and perceived strength and effectiveness. Scores range from 1 to 5 with higher scores indicating greater strength (effect from smoking cigarettes/vaping e-cigarettes) or liking (liking of effect from smoking cigarettes/vaping e-cigarettes)
Minnesota Nicotine Withdrawal Scale (MNWS)(Study 1) | Study visits 2 through 9
  Asses Nicotine withdrawal and smoking craving, anger/irritability, anxiety, depressed mood, restlessness/difficulty concentrating, increased appetite, sleep problems, and somatic symptoms (nausea, constipation, sore throat, dizziness, coughing). Scores range from 0 to 4 with higher scores indicating greater levels of withdrawal (MNWS) or more craving to smoke (MNWS Craving).
Puffing topography: Puff count (Study1) | 60 minute puffing session at each of the 8 study lab visits
  Puff count will be measured.
Puffing topography: Average puff duration (Study1) | 60 minute puffing session at each of the 8 study lab visits
  Average puff duration will be measured.
Puffing topography: inter-puff interval (Study1) | 60 minute puffing session at each of the 8 study lab visits
  Inter-puff interval will be measured.
Puffing topography: Flow rate (Study1) | 60 minute puffing session at each of the 8 study lab visits
  Flow rate will be measured.
Puffing topography: Volume (Study1) | 60 minute puffing session at each of the 8 study lab visits
  Puff volume will be measured.
General Labeled Magnitude Scale (gLMS) (Study 2) | 1 six hour lab visit
  Complete the General Labeled Magnitude Scale (gLMS) after each condition. Scores range from 0 "No Sensation" to 100 "Strongest Imaginable".
Labeled Hedonic Scale (LHS) (Study 2) | 1 six hour lab visit
  Complete the Labeled Hedonic Scale (LHS) after each condition. Scores range from -100 "Most Disliked Imaginable" to 100 "Most Liked Imaginable".
Sensory Attributes (Study 2) | 1 six hour lab visit
  Rate sensory attributes (smoothness, harshness, sweetness, bitterness) on a 100-unit visual analog scale after each condition.
Overall acceptance: Industry-designed Thermometer Rating Scale (Study 2) | 1 six hour lab visit
  Complete a tobacco industry-designed thermometer rating scale of overall acceptance after each condition. Ratings range from 0 "the very worst" to 100 "the very best", with 50 indicating "indifferent".

CONTACTS AND LOCATIONS:
Overall Officials: Theodore L Wagener, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States